CLINICAL TRIAL: NCT00473538
Title: Effects of Structured Exercise Program Versus Hypocaloric Hyperproteic Diet on the Reproductive Function in Obese Anovulatory Infertile Patients With Polycystic Ovary Syndrome: a 24-Week Prospective Study.
Brief Title: Structured Exercise Training Program Versus Hypocaloric Hyperproteic Diet in Obese Anovulatory Infertile Patients With PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01/2004
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2007-11

CONDITIONS: Polycystic Ovary Syndrome; Anovulation; Infertility
Keywords: Structured exercise training program; Infertility; Menstrual cycle; PCOS; Treatment
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anovulation; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Structured exercise training
Behavioral: Hypocaloric hyperproteic diet

SUMMARY:
Lifestyle modifications are successfully employed in polycystic ovarian syndrome (PCOS) improving menstrual cycles and fertility. Unfortunately, the compliance over the time is very low. Recently, we have showed a high adherence to structured exercise training (SET) program in women with PCOS. The current study will be aimed to compare the efficacy of the SET program with a diet program on the reproductive function in obese anovulatory infertile PCOS patients.

DETAILED DESCRIPTION:
Forty obese anovulatory infertile PCOS patients who wish to conceive will be allocated in two study-groups according to their desire: structured exercise training (SET) group (n. 20) will undergo a SET program, whereas diet group (n. 20) will undertake a hypocaloric hyperproteic diet. The duration of the study will be of 24 weeks. At baseline, after 12 and 24 weeks clinical, endocrine and metabolic evaluations will be performed in each patient and all reproductive events obtained throughout the study will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* PCOS
* Anovulatory infertility
* Obesity (BMI >30)

Exclusion Criteria:

* Age <18 or >35 years
* Neoplastic, metabolic, hepatic, renal, and cardiovascular disorders or other concurrent medical illnesses
* Hypothyroidism, hyperprolactinemia, Cushing's syndrome, and non-classical congenital adrenal hyperplasia
* Current or previous (within the last six months) use of oral contraceptives, glucocorticoids, antiandrogens, ovulation induction agents, antidiabetic and anti-obesity drugs or other drugs know to affect sex hormone levels, carbohydrate metabolism, or appetite
* Organic pelvic diseases, previous pelvic surgery, suspected peritoneal factor infertility, tubal or male factor infertility or sub-fertility

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2004-01; Study Completion 2006-08

PRIMARY OUTCOMES:
Pregnancy rate | six months

SECONDARY OUTCOMES:
Menstrual frequency | six months
Abortion rate | six months
Compliance | six months

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, MD, Principal Investigator — Department of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro; Francesco Orio, MD, Principal Investigator — Department of Molecular and Clinical Endocrinology and Oncology, University "Federico II" of Naples, and Chair of Endocrinology, University "Parthenope", of Naples
Locations (1):
- "Pugliese" Hospital, Catanzaro, Italy

REFERENCES:
- [Background] Vigorito C, Giallauria F, Palomba S, Cascella T, Manguso F, Lucci R, De Lorenzo A, Tafuri D, Lombardi G, Colao A, Orio F. Beneficial effects of a three-month structured exercise training program on cardiopulmonary functional capacity in young women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2007 Apr;92(4):1379-84. doi: 10.1210/jc.2006-2794. Epub 2007 Jan 30. PMID 17264174
- [Background] Clark AM, Ledger W, Galletly C, Tomlinson L, Blaney F, Wang X, Norman RJ. Weight loss results in significant improvement in pregnancy and ovulation rates in anovulatory obese women. Hum Reprod. 1995 Oct;10(10):2705-12. doi: 10.1093/oxfordjournals.humrep.a135772. PMID 8567797
- [Background] Norman RJ, Noakes M, Wu R, Davies MJ, Moran L, Wang JX. Improving reproductive performance in overweight/obese women with effective weight management. Hum Reprod Update. 2004 May-Jun;10(3):267-80. doi: 10.1093/humupd/dmh018. PMID 15140873
- [Derived] Palomba S, Giallauria F, Falbo A, Russo T, Oppedisano R, Tolino A, Colao A, Vigorito C, Zullo F, Orio F. Structured exercise training programme versus hypocaloric hyperproteic diet in obese polycystic ovary syndrome patients with anovulatory infertility: a 24-week pilot study. Hum Reprod. 2008 Mar;23(3):642-50. doi: 10.1093/humrep/dem391. Epub 2007 Dec 23. PMID 18158291